CLINICAL TRIAL: NCT02803190
Title: Osteoporosis and Fall Prevention and Posture Correction Interventions in the Metropolitan Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taiwanese Osteoposis Association, Wang Jhan-Yang Charitable Trust Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201604037RINB
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis Fracture
Keywords: Spine curve; Posture; Fracture; sarcopenia; Exercise
MeSH Terms: conditions — Osteoporotic Fractures; Fractures, Bone; Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICG- integrated care group (Experimental): Integraded Care Group
  Interventions: Behavioral: ICG
- MTG- muscle training group (Experimental): Muscle Traing Group
  Interventions: Behavioral: MTG

INTERVENTIONS:
Behavioral: ICG — All participants received a CD-ROM and one hour education on osteoporosis, sarcopenia, frailty, fall prevention, nutrition, low back pain, good posture, and coping strategy and another hour of professional led exercise program with focus on central muscle groups. ICG subjects received once weekly group exercise.
  Arms: ICG- integrated care group
Behavioral: MTG — All participants received a CD-ROM and one hour education on osteoporosis, sarcopenia, frailty, fall prevention, nutrition, low back pain, good posture, and coping strategy and another hour of professional led exercise program on central muscle groups. MTG subjects received twice weekly machine-based resistance training on major and central muscle groups.
  Arms: MTG- muscle training group

SUMMARY:
The investigators' previous studies in 2014 and 2015 have demonstrated that among community-dwelling older adults with high osteoporotic fracture risks. many sarcopenia indices can be improved and bone mineral density (BMD) maintained with different exercise programs. In 2016, the investigators aim to determine the effects of 2 exercise interventions on posture corrections and further improvement of sarcopenic indices

DETAILED DESCRIPTION:
The current study enrolled subjects who already participated in the 2015 study (n=109) at the National Taiwan University Hospital Bei-Hu Branch (NTUHBB). Subjects will be maintained in their original integrated care group (ICG, target n=50) and muscle training group (MTG, target n=50) when possible. If target sample size is not reached, clinic patients are screened for high risk of fall, osteoporosis/fracture by standardized questionnaires or FRAX for enrollments. New participants are randomized into the ICG and MTG groups. Other than assessments provided in 2015, digital photography on posture and low back pain assessments are done in 2016. All participants received a CD-ROM and one hour education on osteoporosis, sarcopenia, frailty, fall prevention, nutrition, low back pain, good posture, and coping strategy and another hour of professional led exercise program with more focus on central muscle groups. ICG subjects received once weekly group exercise while MTG subjects received twice weekly machine-based resistance training on major muscle groups. Major outcomes were muscle mass (measured by bio-impedance analysis), grip strength, walking speed, and lower leg extension power, Chinese version of Oswestry Disability Index v 2.1 score (for low back pain), and spine curve angle (by photography) at baseline and after 12-weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. older than 50 years of age
2. high risk as defined from one of the following criteria: score≥1 on one minute osteoporosis risk questionnaire; 10 year predicted fracture risk≥20% for major osteoporotic fracture or ≥3% for hip fracture from FRAX; fall≥2 times in pass 1 year
3. having a bone mineral density test within one year period
4. having the capability to understand the study and complete the study interventions
5. willing to participate for the intervention and study follow ups

Exclusion Criteria:

1. People younger than 50 years of age
2. Could not communicate because of hearing, visual, or cognitive problems
3. Unable to stand and walk unaided (walking aids are acceptable)

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Lower extremety extensor power | baseline and 12 weeks
  Lower extremity extensor power is measured by isokinetic resistance equipment by a tranined research assistant with standarized protocol.
  We will compare the statistical properties between baseline and after 12 weeks intervention.

SECONDARY OUTCOMES:
appendicular skeletal muscle index | baseline and 12 weeks
  Measured by bioimpedence analysis machine, before and after intervention. We will compare the statistical properties between baseline and after 12 weeks intervention.
grip strength | baseline and 12 weeks
  Measured by dynamometer, before and after intervention. We will compare the statistical properties of between baseline and after 12 weeks intervention.
walking speed | baseline and 12 weeks
  Measured before and after intervention. Subjects are asked to walk 9 meters. The time between 2 and 7 meter mark are recorded. Walking speed is defined as meter/sec We will compare the statistical properties between baseline and after 12 weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No